CLINICAL TRIAL: NCT00023829
Title: Phase III Randomized Study of Adjuvant Therapy for High Risk pT3N0 Prostate Cancer
Brief Title: Adjuvant Radiation Therapy Plus Hormone Therapy Compared With Radiation Therapy Alone in Treating Patients With Stage II or Stage III Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-P-0011; CDR0000068868; CAN-NCIC-PR9
Record Dates: First submitted 2001-09-13; First posted 2003-01-27 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2013-11

CONDITIONS: Prostate Cancer
Keywords: stage III prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide; Flutamide; Chemotherapy, Adjuvant; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- LH-RH agonist plus radiation therapy (Experimental): Luteinizing hormone-releasing hormone (LH-RH) agonist x 2 years plus radiation therapy (RT) to 63.0 - 66.6 Gy
  Interventions: Drug: bicalutamide; Drug: flutamide; Drug: releasing hormone agonist therapy; Procedure: adjuvant therapy; Radiation: radiation therapy
- Radiation therapy alone (Active Comparator): Radiation therapy alone to 63.0 - 66.6 Gy
  Interventions: Procedure: adjuvant therapy; Radiation: radiation therapy
- LH-RH agonist alone (Active Comparator): Luteinizing hormone-releasing hormone (LH-RH) agonist x 2 years
  Interventions: Drug: bicalutamide; Drug: flutamide; Drug: releasing hormone agonist therapy; Procedure: adjuvant therapy

INTERVENTIONS:
Drug: bicalutamide
  Arms: LH-RH agonist alone; LH-RH agonist plus radiation therapy
Drug: flutamide
  Arms: LH-RH agonist alone; LH-RH agonist plus radiation therapy
Drug: releasing hormone agonist therapy
  Arms: LH-RH agonist alone; LH-RH agonist plus radiation therapy
Procedure: adjuvant therapy
Radiation: radiation therapy
  Arms: LH-RH agonist plus radiation therapy; Radiation therapy alone

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Androgens can stimulate the growth of prostate cancer cells. Drugs such as, flutamide or bicalutamide may stop the adrenal glands from producing androgens. Giving radiation therapy with hormone therapy after surgery to remove the tumor may kill any tumor cells remaining after surgery and be an effective treatment for stage II or stage III prostate cancer. It is not yet known if radiation therapy combined with hormone therapy is more effective than either radiation therapy alone or hormone therapy alone in treating stage II or stage III prostate cancer. (Hormone therapy alone group closed as of 12/9/2002.)

PURPOSE: Randomized phase III trial to compare the effectiveness of adjuvant radiation therapy plus hormone therapy to that of radiation therapy alone or hormone therapy alone in treating patients who have stage II or stage III prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall survival, disease-free survival, freedom from distant metastases, and freedom from PSA failure in patients with high-risk stage II or III prostate cancer treated in the adjuvant setting with radiotherapy and hormonal therapy vs radiotherapy alone.
* Compare the qualitative and quantitative toxic effects of these regimens in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to seminal vesicle invasion (yes vs no), preoperative PSA (10 ng/mL or less vs greater than 10 ng/mL), Gleason score (2-6 vs 7 vs 8-10), positive surgical margins (yes vs no), and neoadjuvant hormonal therapy (yes vs no). Patients are randomized to 1 of 3 treatment arms. (Arm III closed to accrual as of 12/9/2002.)

* Arm I: Patients undergo radiotherapy once daily 5 days a week for 7 weeks. Beginning the first day of radiotherapy, patients also receive hormonal therapy comprising a luteinizing-hormone-releasing hormone agonist once every 1-4 months for 2 years AND oral flutamide 3 times daily OR oral bicalutamide once daily for 1 month.
* Arm II: Patients undergo radiotherapy as in arm I.
* Arm III (Closed to accrual as of 12/9/2002):Patients receive hormonal therapy as in arm I.

Patients are followed every 3 months for 1 year, every 6 months for 4 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 1,398 patients (699 per treatment arm) will be accrued for this study within 5 years. (Arm III closed to accrual as of 12/9/2002.)

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed prostate cancer

  * T2-3, N0, M0
  * No metastatic disease
* High-risk for PSA relapse as defined by Gleason score 7 or higher and ≥ 1 of the following OR Gleason score < 7 and ≥ 2 of the following:

  * Preoperative PSA > 10 ng/mL
  * Positive surgical margins
  * Seminal vesicle invasion
* Preoperative PSA ≤ 40.0 ng/mL
* Postoperative PSA ≤ 0.2 ng/mL
* Negative lymph node status by lymph node sampling or dissection

  * If lymph node status is unknown, must have < 5% risk of involvement by Roach formula

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* Zubrod 0-1

Life expectancy:

* Not specified

Hematopoietic:

* WBC ≥ 3,000/mm^3
* Platelet count ≥ 130,000/mm^3
* Hemoglobin ≥ 11.4 g/dL

Hepatic:

* ALT ≤ 3 times normal

Renal:

* Creatinine ≤ 2.5 mg/dL

Other:

* No other prior or concurrent invasive malignancy within the past 5 years except superficial nonmelanoma skin cancer
* No other major medical or psychiatric illness that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 5 years since prior chemotherapy

Endocrine therapy:

* At least 60 days since prior finasteride
* At least 90 days since prior testosterone
* Prior pharmacologic androgen ablation for prostate cancer allowed if initiated within the past 10 months (must switch to study ablation therapy OR discontinue therapy if randomized to receive radiotherapy only)

Radiotherapy:

* No prior radiotherapy to the pelvis
* No concurrent intensity-modulated radiotherapy

Surgery:

* No prior orchiectomy

Ages: 0 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2001-08; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Overall survival | From the date of randomization to the date of death due to any cause

SECONDARY OUTCOMES:
Disease-Free Survival | From the date of randomization to the date of first documented local progression or distant failure
Distant Failure | From the date of randomization to the date of frist documented metastatic disease
Biochemical Failure (detectable PSA) | From the date of randomization to the date of developing a PSA of 0.5 ng/ml or greater over the entry PSA

CONTACTS AND LOCATIONS:
Overall Officials: Richard K. Valicenti, MD, Study Chair — Sidney Kimmel Cancer Center at Thomas Jefferson University; Richard Choo, MD, Study Chair — Toronto Sunnybrook Regional Cancer Centre
Locations (1):
- Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario, Canada